CLINICAL TRIAL: NCT06392672
Title: Evaluation of the Effect of Management of Drug-Related Problems on Clinical Outcomes of Pulmonary Embolism Outpatients
Brief Title: Evaluation of the Effect of Drug-Related Problems in Pulmonary Embolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Istanbul Sultanbeyli State Hospital (Other Government); Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Muhammed Yunus BEKTAY, Dr., Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pahrm. Role in Pulm. Embolism
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Thromboembolisms
Keywords: Pulmonary embolism; bleeding; clinical pharmacist; drug-related problems; anticoagulation
MeSH Terms: conditions — Pulmonary Embolism; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Group: Group in which only observation is made by the clinical pharmacist For patients in this group, no intervention (i.e. recommendation) will be made to physicians by the clinical pharmacist. Within the intervention group, patient characteristics such as the underlying conditions, and the appropriateness of prescribed medications were evaluated for the patients who received treatment for pulmonary embolism and met the inclusion criteria. The participant will take standard treatment. Evaluations will be recorded.
- Intervention Group (Experimental): Intervention Group: Group to which the clinical pharmacist makes recommendations For patients in this group, intervention (i.e. recommendation) will be made to physician in charge by the clinical pharmacist. Within the intervention group, patient characteristics such as the underlying conditions, and the appropriateness of prescribed medications were evaluated for the patients who received treatment for pulmonary embolism and met the inclusion criteria. Through medication reviews, evaluations were made to identify drug-related problems and provide solutions to these problems. The clinical pharmacist provided recommendations to the physicians regarding significant clinically important problems.
  Interventions: Behavioral: Intervention Group: Group to which the clinical pharmacist makes recommendations

INTERVENTIONS:
Behavioral: Intervention Group: Group to which the clinical pharmacist makes recommendations — The drugs administered to patients during scheduled hospital visits will be recorded. A detailed medication review will be conducted by the clinical pharmacist. As a result of a comprehensive evaluation, recommendations were made to doctors regarding drug-related problems and were recorded.
  Arms: Intervention Group

SUMMARY:
Pulmonary embolism (PE) presents notable risks of morbidity and mortality, underscoring the need for customized anticoagulant treatment. There is a scarcity of research examining drug-related issues (DRPs) in PE. This research endeavor seeks to assess how addressing DRPs affects the clinical outcomes of PE patients receiving outpatient care, offering valuable insights to bolster patient safety measures.

This study will conduct a randomized controlled trial on PE patients in Istanbul, Turkey, from January 15, 2022, to January 15, 2023. The intervention group (IG) will receive clinical pharmacist (CP) recommendations for DRPs, while the control group (CG) will undergo observation only. Evaluations will occur at 90- and 180-days post-discharge, focusing on DRPs, CP interventions, and patient outcomes. Data will be systematically recorded and analyzed, adhering to ethical standards and employing the PCNE v9.1 classification system.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) involves the blockage of the pulmonary artery or one of its branches by materials like thrombus from elsewhere in the body. This condition is linked to increased mortality and morbidity rates, and if left untreated, it can result in recurring episodes. Additionally, using anticoagulant therapy poses a significant risk of severe bleeding.

Recent guidelines recommend customizing the duration of PE treatment based on the type of underlying risk factor, distinguishing between transient and persistent factors. Prolonged treatment without a persistent risk factor may heighten the risk of bleeding. Hence, selecting appropriate treatment options tailored to individual patient needs is crucial.

The main goal of our study is to evaluate how managing drug-related problems (DRPs) in pulmonary embolism (PE) outpatients influences their clinical outcomes. This research aims to provide valuable insights into the effectiveness of interventions targeting DRPs within the framework of PE management .

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of pulmonary embolism (ICD-10 code: I26.0)
2. Patients visited the chest diseases outpatient clinic for post-discharge follow-up
3. Being 18 years or older.
4. Patients who could be evaluated by the clinical pharmacist for at least 24 hours within the intervention group.

Exclusion Criteria:

1. Being under 18 years old.
2. Lost follow up in 90th day after pulmonary embolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Acceptance rate of suggested intervention (number) | From the date of randomization until there are 50 patient participants in each group. Average 1 year.
  Acceptance rate of suggested intervention. Dru-related problems and recommendations are classified according to PCNE (Pharmaceutical Care Network Europe) version 9.1. It was recorded how many suggestions were made in the intervention group and how many of these suggestions were accepted.
Bleeding | From the date of randomization until there are 50 patient participants in each group. Average 1 year.
  Occasions of bleeding within the 180th day.

SECONDARY OUTCOMES:
Increase in pulmonary embolism related quality of life | From the date of randomization until there are 50 patient participants in each group. Average 1 year.
  Pulmonary embolism related Quality of life will be assesed after Clinical pharmacist intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)